CLINICAL TRIAL: NCT05541614
Title: Flapless Application of Enamel Matrix Derivative in Class II Mandibular Furcation Defects: a Randomized Clinical Trial
Brief Title: Flapless Application of Enamel Matrix Derivative in Class II Mandibular Furcation Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Georgios Chatzopoulos, PhD candidate, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 155/14-03-2022
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Periodontal Diseases; Periodontal Disease, AVDC Stage 3; Periodontal Disease, AVDC Stage 4; Furcation Defects
Keywords: Periodontal disease; Enamel Matrix Derivative; EMD; Flapless; MINST; Periodontal treatment; Furcation defect
MeSH Terms: conditions — Periodontal Diseases; Furcation Defects

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated at a 1:1 ratio to either subgingival debridement and flapless application of EMD (test group) into the affected furcation defect or to periodontal surgery in combination with EMD application (control group). The selected sites will be randomly assigned to test and control groups using an online software for randomization. The therapist will be kept unaware of treatment allocation until the treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: The selected sites will be randomly assigned to test and control groups using an online software for randomization. The therapist will be kept unaware of treatment allocation until the treatment. The outcomes assessor will be unaware of the treatment allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subgingival debridement + Flapless Enamel Matrix Derivative (Experimental): Subgingival debridement following a minimally-invasive non-surgical treatment (MINST) approach with flapless application of EMD
  Root instrumentation under local anesthesia using mini hand instruments (mini curettes) and ultrasonic instruments with fine tips in the furcation area of mandibular first or second molars with class II buccal furcation defects. EDTA gel will be applied for 2 minutes on the affected root surfaces, followed by rinsing with saline and drying prior to the application of Emdogain® FL. Emdogain® FL has been shown to enhance the early healing of periodontal soft tissue wounds resulting from the instrumentation of periodontal pockets.
  Interventions: Other: Emdogain® FL (flapless Emdogain®) - Enamel Matrix Derivative
- Periodontal surgery + Enamel Matrix Derivative (Active Comparator): Periodontal surgery following a minimally-invasive surgical treatment (MIST) protocol with application of EMD
  Following local anesthesia, minimal flap elevation on the buccal aspect of first or second molars associated with a grade II furcation defect will be performed.Removal of granulation tissues and root instrumentation with mini hand instruments (mini curettes) and ultrasonic instruments with fine tips in the furcation area will then be carried out. EDTA gel will be applied for 2 minutes on the affected root surfaces, followed by rinsing with saline and drying prior to the application of Emdogain®. Then, the surgical flaps will be positioned and sutured in order to completely cover the defects.
  Interventions: Other: Emdogain® - Enamel Matrix Derivative

INTERVENTIONS:
Other: Emdogain® FL (flapless Emdogain®) - Enamel Matrix Derivative — Emdogain® FL has been shown to enhance the early healing of periodontal soft tissue wounds resulting from the instrumentation of periodontal pockets.
  Arms: Subgingival debridement + Flapless Enamel Matrix Derivative
Other: Emdogain® - Enamel Matrix Derivative — Enamel matrix derivative (EMD) has been widely used in the surgical treatment of periodontal disease and in furcation defects.
  Arms: Periodontal surgery + Enamel Matrix Derivative

SUMMARY:
Patients diagnosed with stage III or IV periodontitis that exhibit mandibular first or second molars with increased periodontal probing depth (PPD > 4 mm) and class II buccal mandibular furcation defects (horizontal probing depth of >= 3 mm ) will be recruited. This study will be a non-inferiority, prospective, randomized, double-blind controlled clinical trial with a parallel design. Patient will be recruited from the clinics of the School of Dentistry at the Aristotle University of Thessaloniki and private dental practices in Thessaloniki, Greece. Initially, non-surgical periodontal treatment will be performed through scaling and root planning in combination with oral hygiene instructions and motivation. The re-evaluation will be performed 4-6 weeks following the treatment and the patients who meet the inclusion criteria will be included in the study. Patients will be randomly allocated at a 1:1 ratio to either subgingival debridement and flapless application of EMD (test group) into the affected furcation defect or to periodontal surgery in combination with EMD application (control group). Periodontal and radiographic parameters, patient reported outcomes, oral cavity measurements and gingival crevicular fluid will be collected before as well as up to 9 months following the treatment.

DETAILED DESCRIPTION:
The first step in periodontal therapy aims to successfully remove supragingival dental biofilm, improve oral hygiene and control potential risk factors. During the second step of treatment, the "cause-related therapy", non-surgical periodontal treatment consisting of subgingival debridement aiming to reduce plaque accumulation, calculus deposits, gingival inflammation, pocket depths is performed,which is effective for gaining attachment level. However, non-surgical periodontal treatment per se rarely translates into periodontal regeneration. In patients with severe periodontal disease residual periodontal pockets may remain after an initial therapy. Furcation defects often do not respond favourably to non-surgical periodontal therapy and are associated with elevated risk of progression. The elimination of these residual periodontal pockets can be achieved at the thirdstep of the treatment by resective or regenerative procedures based on the morphology of the defect or alternatively repeated subgingival instrumentation with or without adjunctive therapies can be carried out. Regeneration of the periodontal tissues includes cementum, periodontal ligament (PDL) and alveolar bone. Currently, several flap designs and biomaterials have been utilized and tested in the literature aiming at periodontal regeneration including bone grafts, bone substitute materials, growth factors, enamel matrix derivative proteins (EMD), guided tissue regeneration or even a combination of these materials. Although the application of EMD in conjunction with non-surgical periodontal treatment has shown a positive effect with evidence of regeneration, its effectiveness remains inconclusive.

Further studies in various disease conditions (intrabony defects, furcation defects, suprabony defects) are needed to confirm the potential benefit of adjunctive EMD application in combination with subgingival debridement (non surgical periodontal therapy). No study to our knowledge has tested the efficacy of flapless application of EMD in the healing of molars with furcation involvement.

Study design: Non-inferiority, double-blind, randomized, controlled clinical trial with parallel design.

Null Hypothesis: The adjunctive flapless use of enamel matrix derivative (EMD) during subgingival debridement in patients diagnosed with Stage III or IV periodontitis that exhibit class II buccal mandibular furcation involvement leads to inferior outcomes in clinical and radiographic as well as in biomarkers in comparison with surgical periodontal treatment with EMD.

Hypothesis: The adjunctive flapless use of enamel matrix derivative (EMD) during subgingival debridement in patients diagnosed with Stage III or IV periodontitis that exhibit class II buccal mandibular furcation involvement results in noninferior/equivalent outcome in clinical and radiographic variables as well as in biomarkers in comparison with surgical periodontal treatment with EMD.

Aim: The aim of this study is to investigate the non-inferiority of the flapless application of enamel matrix derivate (EMD) in addition to subgingival debridement in class II buccal mandibular furcationsin regards to the clinical and radiographic outcome as well as the level of biomarkers related to periodontal disease activity, inflammation and regeneration compared with periodontal surgery with EMD.

Methods: Patients diagnosed with stage III or IV periodontitis that exhibit mandibular first or second molars with increased periodontal probing depth (PPD > 4 mm) and class II buccal mandibular furcation defects (horizontal probing depth of >= 3 mm)will be recruited. This study will be a non-inferiority, prospective, randomized, double-blind controlled clinical trial with a parallel design.

Patient will be recruited from the clinics of the School of Dentistry at the Aristotle University of Thessaloniki and private dental practices in Thessaloniki, Greece.

Pre-treatment: Non-surgical periodontal treatment will be performed through scaling and root planning in combination with oral hygiene instructions and motivation. The reevaluation will be performed 4-6 weeks following the treatment and the patients who meet the inclusion criteria will be included in the study. Patients will be randomly allocated at a 1:1 ratio to either subgingival debridement and flapless application of EMD (test group) into the affected furcation defect or to periodontal surgery in combination with EMD application (control group). Periodontal and radiographic parameters, patient reported outcomes, oral cavity measurements and gingival crevicular fluid will be collected before as well as up to 9 months following the treatment.

Sample size calculation An estimate of the expected PPD reduction from OFD+EDTA+EMD was drawn from Casarin et al. 2010. The mean PPD reduction following OFD+EDTA+EMD was 1.9 +/- 1.6 mm and 1.0 +/-1.3 mm when OFD+EDTA was only performed. The differential effect of using EMD in a surgical periodontal treatment amounts about 1 mm. The sample size calculation was performed using α=0.05 and 90% power to detect a difference of 1 mm between treatment groups (MINST+Flapless EMD vs MIST+EMD) which is clinically significant and detectable. The estimated standard deviation was 1 mm. The required sample size was calculated to be 18 individuals in each group (total 36). Considering that some patients might be lost during the follow-up, a total of 44 participants will be enrolled (dropout rate of 20%). When the power was set to 80%, the required sample size is 13 patients per group (total 26). Considering a dropout rate of 20%, a total of 32 patients will be enrolled.

Statistical methods Descriptive statistics will be used to present the results of the sample's characteristics (mean and standard deviation for age, number of teeth, clinical periodontal and radiographic parameters; counts and percentages for categorical variables such as gender, medical and smoking history etc). The distribution of the sample will be measured with the Shapiro-Wilk test. In case of normal distribution: paired and unpaired t-tests will be utilized. In case a non-parametric test is used, Wilcoxon signed-rank and Mann Whitney U tests will be utilized. Chi-square test will be also used to compare categorical variables. GCF and periodontal measurements can be correlated with Spearman or Pearson rank correlation test. A statistical significant result will be set to a threshold level of <=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of at least 18 years of age with a diagnosis of stage III or IV periodontitis.
* Have at least one class II furcation defect with PPD >4 mm and horizontal probing depth of >= 3 mm in a mandibular first or second molar.
* Teeth have to be vital or properly treated endodontically.
* Gingival recession ≤ 2mm on furcation site
* Proper oral hygiene: full-mouth plaque score (FMPS) ≤20%.
* Systemically healthy (absence of systemic conditions such as diabetes mellitus that can affect the treatment outcome of periodontal therapy)
* Ability to understand the study procedures and comply with them through the length of the study.
* Given written informed consent form for participation in the study.

Exclusion Criteria:

* Pregnant or lactating female (self-reported).
* Current acute infection.
* Non-surgical periodontal treatment within the last 6 months or/and surgical periodontal treatment the last 12 months before the initial pre-treatment.
* Need for antibiotic premedication.
* Antibiotic treatment in the previous 3 months.
* Allergy to any materials or medications that could be used during or after the procedure.
* Teeth having an improper endodontic therapy with clinical signs of infection or subgingival restorations.
* Tooth mobility of 2nd and 3rd degree.
* History of radiation therapy in the head and neck region.
* Chronic use of medications that may alter the response of periodontal tissues.
* Smoke ≥ 10 cigarettes/day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Periodontal probing pocket depth (PPD) change | 9 months after treatment
  Changes in pocket probing depth will be measured using a periodontal probe. The depth of the sulcus will be assessed by gently inserting a graduated periodontal probe until resistance is encountered at the base of the sulcus. The depth from the free gingival margin to the base of the sulcus is measured in millimeters and represents PPD.

SECONDARY OUTCOMES:
Horizontal and vertical furcation involvement change. | 9 months after treatment
  Changes in horizontal and vertical furcation involvement will be measured using a periodontal probe.
Periodontal clinical attachment level (CAL) change. | 9 months after treatment
  Changes in clinical attachment level will be measured using a periodontal probe.
Bleeding on Probing (BOP) change | 9 months after treatment
  Bleeding on Probing will be tested using a periodontal probe that is carefully introduced to the bottom of the pocket gently.
Gingival recession (REC) change | 9 months after treatment
  Changes in gingival recession will be measured using a periodontal probe.
Furcation involvement grade change | 9 months after treatment
  Proportion of sites demonstrating change in furcation grade level as measured with Nabers probe
Radiographic defect depth, height, root trunk and width. | 9 months after treatment
  Assessment of the defect depth, height, root trunk and width using Cone-beam computed tomography systems (CBCT) and periapical radiographs and subtraction radiography
Levels of markers related to periodontal disease activity, inflammation as well as regeneration in the GCF. | 9 months after treatment
  The levels of markers will be assessed using gingival crevicular fluid (GCF) and analyzed with multiplex assays (in pg or ng based on the assays)
Patient-reported outcome measures | 9 months after treatment
  Patient-reported outcome measures using Visual Analogue Scales (VAS) Visual analogue Scale: range from 0 mm "no", to 100 mm," the worst possible"
Oral health-related quality of life | 9 months after treatment
  Oral health-related quality of life measures using OHIP-14 (Greek version) The OHIP-14 captures seven domains of OHRQoL with two items per domain: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap.
  The responses are rated on a 5-point Likert scale: 0 = never; 1 = hardly ever; 2 = occasionally; 3 = fairly often; 4 = very often/every day. The OHIP-14 scores can range from 0 to 56 and are calculated by summing the ordinal values for the 14 items.

CONTACTS AND LOCATIONS:
Locations (1):
- Aristotle University of Thessaloniki, School of Dentistry, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] - Graziani F, Karapetsa D, Mardas N, Leow N, Donos N (2018) Surgical treatment of the residual periodontal pocket. Periodontol 2000 76:150-163. - Lang NP, Salvi GE, Sculean A (2019) Nonsurgical therapy for teeth and implants-When and why? Periodontol 200079(1):15-21. doi: 10.1111/prd.12240. - Kaldahl WB, Kalkwarf KL, Patil KD, Molvar MP. Responses of four tooth and site groupings to periodontal therapy. J Periodontol. 1990 Mar;61(3):173-9. doi: 10.1902/jop.1990.61.3.173. PMID: 2181110. - Tomasi C, Leyland AH, Wennström JL. Factors influencing the outcome of non-surgical periodontal treatment: a multilevel approach. J Clin Periodontol. 2007 Aug;34(8):682-90. doi: 10.1111/j.1600-051X.2007.01111.x. PMID: 17635246. - Wang HL, Burgett FG, Shyr Y, Ramfjord S. The influence of molar furcation involvement and mobility on future clinical periodontal attachment loss. J Periodontol. 1994 Jan;65(1):25-9. doi: 10.1902/jop.1994.65.1.25. PMID: 8133412. - Nibali L, Zavattini A, Nagata K, Di Iorio A, Lin GH, Needleman I, Donos N. Tooth loss in molars with and without furcation involvement - a systematic review and meta-analysis. J Clin Periodontol. 2016 Feb;43(2):156-66. doi: 10.1111/jcpe.12497. Epub 2016 Feb 12. PMID: 26932323. - Meza Mauricio J, Furquim CP, Bustillos-Torrez W, Soto-Peñaloza D, Peñarrocha-Oltra D, Retamal- Valdes B, Faveri M (2021) Does enamel matrix derivative application provide additional clinical benefits in the treatment of maxillary Miller class I and II gingival recession? A systematic review and meta-analysis. Clin Oral Investig25(4):1613-1626. doi: 10.1007/s00784-021-03782-2. - Graziani F, Gennai S, Cei S, Ducci F, Discepoli N, Carmignani A, Tonetti M (2014) Does enamel matrix derivative application provide additional clinical benefits in residual periodontal pockets associated with suprabony defects? A systematic review and meta-analysis of randomized clinical trials. J Clin Periodontol;41(4):377-86. doi: 10.1111/jcpe.12218. - Stavropoulos A, Bertl K, Spineli LM, Sculean A, Cortellini P, Tonetti M (2021) Medium- and longterm clinical benefits of periodontal regenerative/reconstructive procedures in intrabony defects: Systematic review and network meta-analysis of randomized controlled clinical studies. J Clin Periodontol48(3):410-430. doi: 10.1111/jcpe.13409. - Esberg A, Isehed C, Holmlund A, Lundberg P (2019) Peri-implant crevicular fluid proteome before and after adjunctive enamel matrix derivative treatment of peri-implantitis. J Clin Periodontol46(6):669-677. doi: 10.1111/jcpe.13108. - Oliveira HFE, Verri F, Lemos CA, Cruz R, Batista VES, Pellizzer E, Santinoni C (2020) Clinical Evidence for Treatment of Class II Periodontal Furcation Defects. Systematic Review and Metaanalysis. J Int Acad Periodontol22(3):117-128. - Wennstrom JL, Lindhe J (2002) Some effects of enamel matrix proteins on wound healing in the dentogingival region. J Clin Periodontol29:9-14. - Mark R, Mohan R, Gundappa M, Balaji MDS, Vijay VK, Umayal M. Comparative Evaluation of Periodontal Osseous Defects Using Direct Digital Radiography and Cone-Beam Computed Tomography. J Pharm Bioallied Sci. 2021 Jun;13(Suppl 1):S306-S311. doi: 10.4103/jpbs.JPBS_804_20. Epub 2021 Jun 5. PMID: 34447099; PMCID: PMC8375921. - Assiri H, Dawasaz AA, Alahmari A, Asiri Z. Cone beam computed tomography (CBCT) in periodontal diseases: a Systematic review based on the efficacy model. BMC Oral Health. 2020 Jul 8;20(1):191. doi: 10.1186/s12903- 020-01106-6. PMID: 32641102; PMCID: PMC7341656. - Walter C, Schmidt JC, Rinne CA, Mendes S, Dula K, Sculean A. Cone beam computed tomography (CBCT) for diagnosis and treatment planning in periodontology: systematic review update. Clin Oral Investig. 2020 Sep;24(9):2943-2958. doi: 10.1007/s00784-020-03326-0. Epub 2020 Jul 3. PMID: 32617781. - Yusof NAM, Noor E, Reduwan NH, Yusof MYPM. Diagnostic accuracy of periapical radiograph, cone beam computed tomography, and intrasurgical linear measurement techniques for assessing furcation defects: a longitudinal randomised controlled trial. Clin Oral Investig. 2021 Mar;25(3):923-932. doi: 10.1007/s00784-020- 03380-8. Epub 2020 Jun 14. PMID: 32535703. - Zhang W, Foss K, Wang BY. A retrospective study on molar furcation assessment via clinical detection, intraoral radiography and cone beam computed tomography. BMC Oral Health. 2018 May 3;18(1):75. doi: 10.1186/s12903- 018-0544-0. PMID: 29724208; PMCID: PMC5934848.